CLINICAL TRIAL: NCT05420090
Title: The Effects of Milk and Banana Given as a Night Meal to Individuals Diagnosed With Sleep Disorders on Sleep Quality, BDNF and Appetite Mechanism
Brief Title: The Effects of Milk and Banana as a Night Meal to Primary Insomnia on Sleep Quality, BDNF and Appetite Mechanism
Acronym: diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2022-06-01; First posted 2022-06-15 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Primary Insomnia
Keywords: diet; food; BDNF; Appetite
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 1. Experimental: Banana arm Experimental: Milk arm Control arm
Who Masked: Investigator
Masking Description: ınvestigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eating banana for 6 weeks before bedtime (Experimental): Participants will consume 1 portion of banana (gross 80-85 g) given to them for 6 weeks, approximately 45 minutes-1 hour before bedtime.
  Interventions: Behavioral: Banana arm
- drinking milk for 6 weeks before bedtime (Experimental): Participants will consume 200 ml of whole milk given to them for 6 weeks, approximately 45 minutes-1 hour before bedtime.
  Interventions: Behavioral: Milk arm
- Control (Experimental): Not making any changes in diet
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Banana arm — Venous blood samples will be taken from the participants in 3 groups before starting the study. Pittsburgh Sleep Quality Index will be applied.Food consumption frequency and food-based follow-up will be carried out.Participants will consume 1 portion of banana (gross 80-85 g) given to them for 6 weeks, approximately 45 minutes-1 hour before bedtime. The frequency of food consumption will be taken from the participants each week.
  Arms: eating banana for 6 weeks before bedtime
Behavioral: Milk arm — Venous blood samples will be taken from the participants in 3 groups before starting the study. Pittsburgh Sleep Quality Index will be applied. Food consumption frequency and food-based follow-up will be carried out. Participants will consume 200 ml of whole milk given to them for 6 weeks, approximately 45 minutes-1 hour before bedtime. The frequency of food consumption will be taken from the participants each week.
  Arms: drinking milk for 6 weeks before bedtime
Behavioral: No intervention — Venous blood samples will be taken from the participants in 3 groups before starting the study. Pittsburgh Sleep Quality Index will be applied. The frequency of food consumption will be taken from the participants each week.Participants are expected not to make any changes in their diet. As in other groups, the frequency of food consumption will be taken from the participants every week in this group. In order to observe the possible changes in the experimental arms, the individuals in the control arm will be asked not to consume bananas and whole milk after 16:00 and they will be informed about this.
  Arms: Control

SUMMARY:
The aim of this study to determine the impact of banana and milk on sleep and appetite

DETAILED DESCRIPTION:
Sleep is one of the main components of the continuity of circadian rhythm. It restores energy and enhancement, memory. Sleep disturbances and short sleep duration are important risk factors for many diseases. Nutrition is one of the main determinants of health status in many diseases related to inflammation. Especially the night meal, known as the foods consumed before bedtime, has a strong effect on sleep. Although there are methodological differences, most studies show that unhealthy eating habits are associated with short sleep duration. It is thought that consuming foods with high tryptophan and melatonin content can reduce sleep problems. This study will give a chance to observe the effects of nutrients on sleep and appetite mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Applying to the Sleep Polyclinic,
* 18-45 years old,
* Body Mass Index (BMI) between 18.5-25 kg/m2,
* Male and female patients diagnosed with primary sleep disorder for the first time

Exclusion Criteria:

* Individuals with any psychiatric illness,
* Those who use cigarettes, alcohol, drugs or sedative drugs,
* Individuals with any chronic disease (diabetes, etc.),
* Pregnant and/or lactating
* Individuals with lactose intolerance,
* athletes,
* Individuals who are allergic to bananas
* Individuals with lactose intolerance or milk intolerance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender homogenity will be based
Enrollment: 21 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Changing Score on the Pittsburgh Sleep Quality Index (PSQI) from baseline | at baseline, 6. week
  Change from baseline PSQI at 6 weeks
Level of Brain Derived Neurotrophic Factor (pg/ml) | at baseline, 6. week
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done (ng/ml)
Level of Leptin (mg/dl) | at baseline, 6. week
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done (ng/ml)
Level of Ghrelin (mg/dl) | at baseline and 6. week
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done (ng/ml))
Evaluate stages of sleep and the oxygen level in blood | at baseline and 6. week
  Polymsomnography is used for the diagnosis and treatment plan of sleep disorder and sleep architecture

SECONDARY OUTCOMES:
Nutrient intake (g/day) | 6 consecutive weeks, 6 weeks
  assessed by a food frequency record as g/day

CONTACTS AND LOCATIONS:
Overall Officials: Muteber Gizem KESER, PhD,Lecturer, Principal Investigator — KTO Karatay University
Locations (1):
- Selcuk University Medical Faculty, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No